CLINICAL TRIAL: NCT00084175
Title: HIV/STD Safer Sex Skills Groups for Men in Drug Treatment Programs
Brief Title: HIV/STD Safer Sex Skills Groups for Men in Drug Treatment Programs - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Donald Calsyn, Ph.D., University of Washington
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTN-0018-1
Record Dates: First submitted 2004-06-08; First posted 2004-06-09 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Behavior Therapy
Keywords: behavioral intervention
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to evaluate a five-session Human Immunodeficiency Virus/Acquired Immune Deficiency Disease (HIV/AIDS) group therapy designed specifically for heterosexual men. This therapy is compared to standard HIV/AIDS education, which generally consists of a single session of HIV education.

ELIGIBILITY:
All adult males age 18 and above in drug abuse treatment at participating Community Treatment Providers will be invited to participate.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630
Dates: Start 2004-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
AIDS risk behavior

CONTACTS AND LOCATIONS:
Overall Officials: Donald Calsyn, Ph.D., Principal Investigator — University of Washington
Locations (14):
- United States (14):
  - Matrix Institute on Addictions, Rancho Cucamonga, California
  - San Francisco General Hospital, San Francisco, California
  - Hartford Dispensary, New Britain, Connecticut
  - CT Renaissance, Inc., Norwalk, Connecticut
  - Life Link, Santa Fe, New Mexico
  - Staten Island University Hospital, Staten Island, New York
  - Addiction Drug Services-Highpoint, High Point, North Carolina
  - South Light, Raleigh, North Carolina
  - Comprehensive Addiction Services System, Toledo, Ohio
  - The Consortium, Philadelphia, Pennsylvania
  - Thomas Jefferson Intensive Sub. Abuse TP, Philadelphia, Pennsylvania
  - LRADAC-Lexington-Richmond Alcohol & Drug Council, Columbia, South Carolina
  - Evergreen Treatment Services, Seattle, Washington
  - Prestera Center for Mental Health Svcs., Huntington, West Virginia

REFERENCES:
- [Derived] Calsyn DA, Campbell AN, Tross S, Hatch-Maillette MA. Is monogamy or committed relationship status a marker for low sexual risk among men in substance abuse treatment? Clinical and methodological considerations. Am J Drug Alcohol Abuse. 2011 Sep;37(5):294-300. doi: 10.3109/00952990.2011.596874. PMID 21854271
- [Derived] Calsyn DA, Crits-Christoph P, Hatch-Maillette MA, Doyle SR, Song YS, Coyer S, Pelta S. Reducing sex under the influence of drugs or alcohol for patients in substance abuse treatment. Addiction. 2010 Jan;105(1):100-8. doi: 10.1111/j.1360-0443.2009.02812.x. PMID 20078464
- [Derived] Calsyn DA, Hatch-Maillette M, Tross S, Doyle SR, Crits-Christoph P, Song YS, Harrer JM, Lalos G, Berns SB. Motivational and skills training HIV/sexually transmitted infection sexual risk reduction groups for men. J Subst Abuse Treat. 2009 Sep;37(2):138-50. doi: 10.1016/j.jsat.2008.11.008. Epub 2009 Jan 15. PMID 19150206